CLINICAL TRIAL: NCT03330587
Title: Living Alone in Old Age With Cognitive Impairment
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: R01AG069147 (NIH)
Record Dates: First submitted 2017-08-24; First posted 2017-11-06 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Living Alone; Alzheimer Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to better understand the experience of living alone in older age with cognitive impairment.

We recruit adults 55+ living alone with cognitive impairment such as Alzheimer's disease or mild cognitive impairment.

This study investigates the priorities and concerns of older adults living alone with cognitive impairment. Participants are interviewed 5 times for one hour in their homes within 3 months at a time that works for them.

DETAILED DESCRIPTION:
The purpose of this study is to better understand the experience of living alone in older age with cognitive impairment. This knowledge is important to design programs that are appropriate. Dr. Elena Portacolone, an Assistant Professor from the Institute of Health and Aging is the study researcher.

Study participants are interviewed by Elena at a time and place convenient to them, usually their home. Interviews are audio recorded and last around one hour. Study participants are interviewed five times within 3 months.

After the interview, a transcriptionist will type into a computer the recording and will remove personal names. The sound recording will then be destroyed.

Participants can stop being in the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Living alone
* Medical diagnosis of Alzheimer's disease or mild cognitive impairment

Exclusion Criteria:

* Living in nursing homes, assistive living facilities.
* Alcohol abuse

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons over 55 years of age living alone and having a medical diagnosis of Alzheimer's disease or mild cognitive impairment
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Ethnographic interviews | One hour
  Questions that follow the train of thought of study participants

CONTACTS AND LOCATIONS:
Overall Officials: Elena Portacolone, PhD MPH MBA, Principal Investigator — University of California, San Francisco
Locations (1):
- Institute for Health & Aging, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The investigator discusses her study — https://www.youtube.com/watch?v=KNbkvlQvxLI